CLINICAL TRIAL: NCT03309215
Title: Evaluation of the Clinical Implication of Short Repeated Nickel Exposures
Brief Title: Short Repeated Nickel Exposures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Malin Glindvad Ahlström, MD, Ph.d.-student, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-16050296; HGH-2017-027 (Other: Data Protection Agency Region Hovedstaden)
Record Dates: First submitted 2017-10-04; First posted 2017-10-13 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Allergic Contact Dermatitis Due to Nickel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with nickel allergy (Experimental): Experimental stimulation with nickel discs
  Interventions: Other: Experimental stimulation with nickel discs
- Persons without nickel allergy (Experimental): Experimental stimulation with nickel discs
  Interventions: Other: Experimental stimulation with nickel discs

INTERVENTIONS:
Other: Experimental stimulation with nickel discs — All participants will be exposed to 8 metal discs, 3 cm in diameter, 4 on each arm, placed on the volar side of the forearms (figure 1). Three of the metallic discs consists of >99 wt.% nickel one consist of >99wt.% Aluminium.The latter is used as a negative control. The discs will be applied under occlusion and with initial pressure and friction.
  One metallic disc with nickel, and one with aluminium, will be randomized for the earlobes on the patients with nickel allergy

SUMMARY:
The former Nickel Directive was introduced in EU in 1994 limiting the release of nickel from items intended for prolonged contact with skin. The nickel regulation entered into full force in 2001 and became a part of REACH (the EU chemicals regulation) in 2009. Since then the prevalence of nickel allergy has declined in some countries, but not in others, following the implementation. Young individuals still become allergic to nickel (2, 3) and a high prevalence of nickel allergy, exceeding 10%, is seen among young women (below 30 years) in the general population.

The EU nickel regulation has been changing over time. The present limits of nickel release for metallic items intended for direct and prolonged contact with the skin is <0.5 μg/cm2/week and <0.2 μg/cm2/week for any post assemblies inserted into pierced holes. In 2014, EU defined prolonged contact with the skin as: at least 30 minutes on one or more occasions within two weeks for items with continuous skin contact, or to at least 10 minutes on three or more occasions within two weeks (7).

The overall objective is to evaluate how well the EU nickel regulation protects individuals against developing nickel dermatitis. More specifically we will:

1. Study the penetration of nickel in normal and irritated skin after short repeated skin exposure under controlled temperature in nickel sensitized patients and in healthy controls
2. Reveal the potential of short repeated nickel skin exposure on normal and irritated skin to elicit dermatitis, during controlled climate factors in nickel sensitized patients and controls using the time restrictions of the definition of prolonged skin contact in the nickel regulation.

ELIGIBILITY:
For patients with nickel allergy:

Inclusion Criteria:

* Positive patch test to nickel sulphate 5% pet. according to European society of contact dermatitis(ESCD) guidelines within the last 5 years at the Department of Dermatology and Allergy, Gentofte Hospital.
* Age 18-75 years.

Exclusion Criteria:

* Active eczema in test areas
* Generalized eczema
* Scar tissue in test areas.
* Pregnancy or breast feeding
* Treatment with topical corticosteroids or other immune-suppressants on/near test areas within four weeks prior to study start
* Systemic immunomodulatory* treatment within 4 weeks prior to study start
* UV exposure of test areas within three weeks prior to study start
* Participation in other clinical studies within four weeks prior to study start
* Unable to cooperate or communicate with the investigators *Systemic immunomodulatory treatment is drugs taken orally or by injection that modify the response of the immune system by increasing (immunostimulators) or decreasing (immunosuppressives) the production of serum antibodies

For Healthy volunteers:

Inclusion Criteria:

* Negative patch test result to nickel sulphate 5% pet. according to ESCD guidelines (48) at the Department of Dermatology and Allergy, Gentofte Hospital
* Age 18-75 years.

Exclusion Criteria:

* History of contact allergy
* Generalized eczema
* Scar tissue in test areas.
* Pregnancy or breast feeding
* Treatment with topical corticosteroids or other immune-suppressants on/near test areas within four weeks prior to study start
* Systemic immunomodulatory treatment within four weeks prior to study start
* UV exposure of test areas within three weeks prior to study start
* Participation in other clinical studies within four weeks prior to study start
* Unable to cooperate or communicate with the investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-16 (Actual); Primary Completion 2017-12-10 (Actual); Study Completion 2017-12-10 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of development of dermatitis after stimulation over time | 24 hours and 78 hours post stimulation with nickel discs
  Development of dermatitis after stimulation with nickel discs as a change from baseline skin assessment. The criteria developed by the International Contact Dermatitis Research Group (ICDRG), later modified by Hindsén and Bruze will be used for assessment
Change of baseline blood flow over time after stimulation | 24 hours and 78 hours post stimulation with nickel discs
  measure blood flow with laser doppler technique as a surrogate for inflammation on skin following stimulation with nickel discs over time
Nickel skin penetration at different time points after stimulation | Immediate deposition and penetration, 24 hours and 78 hours post stimulation of nickel discs
  by using the tape stripping technique we will measure the deposition of nickel and the penetration of nickel in the stratum corneum following stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Malin G Ahlström, MD, Principal Investigator — National Allergy Research Centre, Department of Allergy and Dermatology
Locations (1):
- Department of Allergy and Dermatology, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Erfani B, Liden C, Midander K. Short and frequent skin contact with nickel. Contact Dermatitis. 2015 Oct;73(4):222-30. doi: 10.1111/cod.12426. Epub 2015 Jun 18. PMID 26086991
- [Result] Hostynek JJ, Dreher F, Nakada T, Schwindt D, Anigbogu A, Maibach HI. Human stratum corneum adsorption of nickel salts. Investigation of depth profiles by tape stripping in vivo. Acta Derm Venereol Suppl (Stockh). 2001;(212):11-8. doi: 10.1080/000155501753279587. PMID 11802472
- [Result] Emilson A, Lindberg M, Forslind B. The temperature effect on in vitro penetration of sodium lauryl sulfate and nickel chloride through human skin. Acta Derm Venereol. 1993 Jun;73(3):203-7. doi: 10.2340/0001555573203207. PMID 8105620
- [Result] Fullerton A, Hoelgaard A. Binding of nickel to human epidermis in vitro. Br J Dermatol. 1988 Nov;119(5):675-82. doi: 10.1111/j.1365-2133.1988.tb03482.x. PMID 3207621
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/3207621
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=The+temperature+effect+on+in+vitro+penetration+of+sodium+lauryl+sulfate+and+nickel+chloride+through+human+skin.+Acta+Derm+Venereol.
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Short+and+frequent+skin+contact+with+nickel
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Human+stratum+corneum+adsorption+of+nickel+salts.+Investigation+of+depth+profiles+by+tape+stripping+in+vivo.